CLINICAL TRIAL: NCT05678894
Title: Single-center Comparative Study of Variation in Acetabular Anteversion According to Pelvic Tilt in Patients With Femoro-acetabular Impingement and Healthy Volunteers.
Acronym: VARIA-CFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A01313-40
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Femoro-acetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- femoro-acetabular impingement (Experimental): symptomatic patients with femoro-acetabular impingement
  Interventions: Other: Scanner and EOS imaging
- Healthy volunteers (Other): Healthy volunteers
  Interventions: Other: Scanner and EOS imaging

INTERVENTIONS:
Other: Scanner and EOS imaging — Cross-sectional imaging and 3D reconstruction to measure and compare acetabular anteversion in 4 functional pelvic positions.

SUMMARY:
The main objective is to show that the upper acetabular anteversions calculated in standing, sitting, sitting hip in maximum flexion and supine positions are lower in patients with symptomatic DWI compared to healthy volunteers.

DETAILED DESCRIPTION:
The study will be presented to a population of symptomatic DWI patients who are offered hip arthroscopy. As these measurements have never been performed before in a control population, the study will also be proposed to a population of healthy volunteers, matched by age, sex, BMI and level of sports activity, in order to have comparative reference values.

The study consisted of cross-sectional imaging and 3D reconstruction to measure and compare acetabular anteversion in 4 functional pelvic positions in both groups.

* Group 1: Symptomatic DWI patients
* Group 2: Healthy volunteers

For symptomatic patients, the preoperative workup will be the same as in routine practice and will include an X-ray as well as a CT scan. Low-dose EOS imaging of the pelvis in profile in 3 positions (standing sagittal tilt, sitting, maximum hip flexion) will complete this workup in the context of the study, to know the sacral slope associated with each of these positions. If the preoperative workup does not include a CT or arthroscan scan with measurement of femoral anteversion, it will be requested in the low-dose protocol.

The control group will perform a CT scan and EOS imaging in the same 3 positions as the patient group.

From the CT scan, a 3D reconstruction with the BoneMetrix software to calculate the superior acetabular anteversion plane will be performed, giving the anteversion for a supine patient. The software also allows to modify the orientation of the pelvis, according to the results of the sacral slope obtained from the EOS assessment for the calculation of the superior acetabular anteversion in the 3 requested positions. Finally, this 3D reconstruction will allow us to search for the impingement dynamically after pelvis-femur segmentation and to measure the position (degree of femoral flexion) in which it occurs.

As these measurements have never been performed before, a control population is needed to obtain reference values for acetabular behavior that does not lead to symptomatic CFA. This population will be matched by age, sex, BMI and sports activity to the study population.

The results obtained from the 2 populations will be compared. For the operated DWI patients in the cohort, the clinical scores will be evaluated at 6 months and 2 years postoperatively to search for a correlation between these scores and the superior acetabular version angles obtained.

This monocentric study will take place at the Clinique de la Sauvegarde. Patients will be seen in consultation by Dr Bonin or Dr Guicherd. They will be included during the pre-operative consultation during which they will be presented with the examinations to be performed, as well as the study. Their consent will be sought before any preliminary procedure. Imaging will be performed at the Clinique du Parc, as is already done for these patients, outside of any study.

ELIGIBILITY:
Inclusion criteria for symptomatic patients:

* Patient at least 18 years of age but < 50 years of age
* Patient with a confirmed diagnosis of DWI for whom arthroscopic impingement surgery is proposed
* Patient who has given and signed free and informed consent
* A patient who is a member of a social security plan or a beneficiary of such a plan

Healthy volunteer inclusion criteria:

* Person at least 18 years of age but < 50 years of age
* Person with no existing DWI diagnosis
* Person who has given and signed free and informed consent
* Person affiliated with a social security plan or beneficiary of such a plan

Exclusion Criteria:

* Patient who has already undergone surgery on the same hip
* Patient with previous spine surgery
* Patient already included in the study for the opposite hip
* Pregnant or breastfeeding patient
* Patient who did not give consent
* Patient for whom it is impossible to give informed information
* Mentally impaired or any other reason that may interfere with understanding
* Patient under court protection, guardianship or curatorship
* Patient in an exclusion period as determined by another study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Anteversions comparison | Day 0
  Comparison of anteversions of the superior plane of the acetabulum obtained from 3D CT reconstruction of the pelvis positioned standing, seated, seated hip in maximum flexion, and supine after matching by low-dose EOS X-ray images, between patients with symptomatic DWI and healthy volunteers.

SECONDARY OUTCOMES:
Functional limitation | Month 6
  Functional limitation, the degree of activity via the HAGOS score
Functional limitation | Month 24
  Functional limitation, the degree of activity via the HAGOS score
Subject quality of life | Month 6
  Quality of life measured by the iHOT questionnaire
Subject quality of life | Month 24
  Quality of life measured by the iHOT questionnaire
Return to previous activities | Month 6
  Return to previous activities measured by mHHS score
Return to previous activities | Month 24
  Return to previous activities measured by mHHS score
Postoperative satisfaction | Month 6
  Postoperative satisfaction measured by the numerical satisfaction scale (ENS)
Postoperative satisfaction | Month 24
  Postoperative satisfaction measured by the numerical satisfaction scale (ENS)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No